CLINICAL TRIAL: NCT01316432
Title: A Study Assessing The Pharmacokinetics, Pharmacodynamics, Safety And Tolerability Of Subcutaneous Bolus And Subcutaneous Infusion Of Cenderitide In Patients With Chronic Heart Failure With Volume Overload (HF)
Brief Title: PK/PD Study of Subcutaneous Cenderitide Infusion in CHF Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nile Therapeutics (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: NIL-CDNP-CT006
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure; ADHF; Chronic Heart Failure; CHF
Keywords: Cenderitide; CD-NP; Natriuretic peptide; Heart failure; Chronic heart failure; HF; CHF
MeSH Terms: conditions — Heart Failure | interventions — cenderitide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- SQ Bolus Cenderitide (Experimental)
  Interventions: Drug: Cenderitide
- SQ Infusion Cenderitide (Experimental): 24 hour SQ infusion of cenderitide
  Interventions: Drug: Cenderitide
- Placebo (Placebo Comparator): 24 hrs of SQ placebo infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cenderitide — Cenderitide is a novel rationally designed chimeric natriuretic peptide to be administered in this trial as either a subcutaneous injection or infusion.
  Other Names: CD-NP
  Arms: SQ Bolus Cenderitide; SQ Infusion Cenderitide
Other: Placebo — Placebo will be administered as a 24-hour SQ infusion
  Arms: Placebo

SUMMARY:
The purposed of the study is to evaluate the pharmacokinetics (PK) response of continuous subcutaneous (SQ) infusion of cenderitide, as compared with a single SQ bolus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Documented systolic heart failure with ejection fraction (EF) ≤ 40%
* Clinical evidence of volume overload
* Systolic blood pressure ≥ 120 mmHg and ≤ 200 mmHg and diastolic blood pressure > 60 mmHg and < 110 mmHg at the time of screening.
* Stable doses of oral medication at least 24 hours prior to screening
* No known allergy or contraindication to furosemide (Lasix®)
* Female patients must be post-menopausal or surgically sterile. A woman may be considered to be surgically sterilized if she has had a bilateral tubal ligation (for at least 6 months), bilateral oophorectomy or complete hysterectomy.
* Be adequately informed of the nature and risks of the study and give written informed consent prior to receiving study medication.

Exclusion Criteria:

* Acute or suspected acute myocardial infarction (AMI) or troponin levels > 5X the upper limit of normal at the institution's local laboratory and accompanied by dynamic ECG changes consistent with AMI
* Clinical diagnosis of acute coronary syndrome (ACS) within 30 days prior to screening.
* Evidence of uncorrected volume or sodium depletion (NA ≤ 130) or other condition that would predispose the patient to adverse events.
* Clinically significant aortic or mitral valve stenosis.
* Temperature > 38°C (oral or equivalent), sepsis or active infection requiring IV anti-microbial treatment.
* ADHF associated with significant arrhythmias (ventricular tachycardia, bradyarrhythmias with ventricular rate < 45 beats per minute or atrial fibrillation/flutter with ventricular response of > 160 beats per minute).
* Severe renal failure defined as creatinine clearance < 30 mL/min as estimated by both the Cockcroft-Gault and the Modification of Diet in Renal Disease (MDRD) equations.
* Significant pulmonary disease (history of oral daily steroid dependency, history of CO2 retention or need for intubation for acute exacerbation, or currently receiving IV steroids).
* Any organ transplant recipient, currently listed (anticipated in the next 60 days) for transplant, or admitted for cardiac transplantation.
* Major surgery within 30 days.
* Major neurologic event, including cerebrovascular events in the prior 60 days.
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral filling patterns).
* Known hepatic impairment
* Received an investigational drug within 30 days prior to screening.
* Women who are pregnant or breastfeeding.
* Known hypersensitivity or allergy to natriuretic peptide or its components, nesiritide, other natriuretic peptides or related compounds.
* Any condition which, in the opinion of the Investigator, could interfere with, or for which the treatment might interfere with the conduct of the study, or which would unacceptably increase the risk of the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) | Up to 36 hours
  Pharmacokinetic measurements of subcutaneous cenderitide infusion compared with a subcutaneous bolus administration

SECONDARY OUTCOMES:
Pharmacodynamics (PD) | Up to 36 hours
  Pharmacodynamics, safey and tolerability will be measured by BP, heart rate, and plasma cGMP after administration.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Orange County Research Center, Tustin, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Analab Clinical Research, Inc., Lenexa, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Hennepin County Medical Center, Minneapolis, Minnesota